CLINICAL TRIAL: NCT01596894
Title: A Randomized, Single Blinded, Controlled, Multi Center Phase 4 Study for Induction of Remission in Active Pediatric Crohn's Disease, Using 2 Months Antibiotic Course of Azithromycin Combined With Metronidazole vs. Metronidazole Alone.
Brief Title: Azithromycin Based Therapy for Induction of Remission in Active Pediatric Crohn's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Prof. Arie Levine (Other Government)
Responsible Party: Sponsor-Investigator, Prof. Arie Levine, Director, Pediatric Gastroenterology and Nutrition unit., Wolfson Medical Center
Organization: Wolfson Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0035-12-WOMC
Record Dates: First submitted 2012-04-12; First posted 2012-05-11 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Crohn's Disease
Keywords: Pediatric; Crohn's disease; Azithromycin; Metronidazole; Mild to moderate Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Azithromycin; Metronidazole

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azithromycin + Metronidazole (Experimental): Oral Azithromycin 7.5 mg/kg once daily (maximum 500mg) 5 consecutive days a week for the first 4 weeks and 3 consecutive days a week for the last 4 weeks +metronidazole 10mg/kg X2/day (maximum 1000mg) for 8 weeks.
  Interventions: Drug: Azithromycin + Metronidazole
- Metronidazole (Active Comparator): Oral metronidazole 10mg/kg X2/day (maximum 1000mg) for 8 weeks.
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: Azithromycin + Metronidazole — Azithromycin 7.5 mg/kg once daily (maximum 500mg) 5 consecutive days a week for the first 4 weeks and 3 consecutive days a week for the next 4 weeks +metronidazole 10mg/kg X2/day (maximum 1000mg) for 8 weeks.
  Other Names: Azanil; Flagyl
  Arms: Azithromycin + Metronidazole
Drug: Metronidazole — Oral metronidazole 10mg/kg X2/day (maximum 1000mg) for 8 weeks.
  Other Names: Flagyl
  Arms: Metronidazole

SUMMARY:
The purpose of this study is to evaluate effectiveness of 2 months antibiotic course of Azithromycin combined with Metronidazole compared with 2 months antibiotic course of Metronidazole alone.

DETAILED DESCRIPTION:
Background: Recent reviews and guidelines no longer recommend antibiotic therapy for induction of remission in Crohn's disease (CD) due to studies showing lack of efficacy. Genetic and microbiological findings have demonstrated that CD is characterized by a defective innate immune response to bacteria and defective apoptosis of T cells. Bacteria have been shown to reside on, and invade epithelial cells, are present in granulomas and to replicate inside macrophage phagolysosomes in susceptible individuals. A defect in bacterial triggering from the luminal epithelial and intracellular compartments, while simultaneously trying to induce apoptosis, has never been explored. Azithromycin is an antibiotic with excellent intracellular penetration, high luminal concentrations, and is also effective against biofilms which have been described in CD. It is a potent activator of apoptosis of T cells. Preliminary data in pediatric patients with short duration of disease have shown a remission rate of 60% and normalization of CRP in about 50% of patients treated with azithromycin and metronidazole in combination. The investigators hypothesize that a 2-month antibiotic course of azithromycin combined with metronidazole is effective for inducing remission in active pediatric Crohns disease (CD). The investigators also hypothesize that remission will be accompanied by normalization of CRP in a high proportion of patients with active CD. The goal of the present study is to evaluate the efficacy of this combination in a randomized controlled trial (RCT).

Methods: This will be a single blinded multicenter randomized controlled trial in children with mild to moderate active CD (PCDAI≥10 ≤40) and elevated CRP, involving the terminal ileum and/or colon , comparing two arms over 8 weeks of therapy:

Group 1: Oral Azithromycin 7.5 mg/kg once daily (maximum 500mg) 5 consecutive days a week for the first 4 weeks and 3 consecutive days a week for the last 4 weeks +metronidazole 10mg/kg X2/day (maximum 1000mg) for 8 weeks .Group 2: Oral metronidazole 10mg/kg X2/day (maximum 1000mg) for 8 weeks . Four visits will take place at enrolment, and at 4, 8, and 12 weeks thereafter. In addition, there will be a telephone visit at 48 hours after commencement of therapy. Patients will be evaluated for PCDAI, Physicians Global Assessment (PGA) and CRP at each visit. The primary endpoint will be response rate at 8 weeks defined as a drop in PCDAI of at least 12.5 points (or remission). Secondary end points will include : 1.Remission rate at 8 weeks. 2. Normalization of CRP (CRP ≤0.5 mg/dL), 3. Fecal calprotectin at 8 weeks and 4. Corticosteroid free remission at 12 weeks.

Importance and anticipated outcomes: The investigators believe that high dose azithromycin will be associated with a high remission rate in early disease. If azithromycin based therapy is validated in an appropriate RCT, it would strengthen the premise that bacteria could, and possibly should be a therapeutic target in CD early in the disease. At a practical level an additional treatment that does not involve corticosteroids and does not suppress the immune system would be available for induction of remission. On a translational level, the underlying hypothesis which led to this treatment regimen, namely that bacteria in all compartments and apoptosis need to be targeted simultaneously, might have ramifications for how the disease should be treated. Theoretically, CD may be a chronic disease because the investigators do not simultaneously treat the two triggers for persistent inflammation (bacterial triggering and defective apoptosis), and ongoing inflammation allows continuous bacterial penetration.

ELIGIBILITY:
Inclusion Criteria:

1. Children 5-17 years of age.
2. Diagnosis of active Crohn's Disease.4. Patients with a PCDAI≥10 ≤40 (mild to moderate disease).
3. Have involvement of the colon and/or terminal ileum.
4. Disease defined as L1, L2, L3 or any of the above and may have gastric, duodenal or esophageal disease (L4a) according to the Paris classification for site of disease.
5. The CRP ≥ 0.6 mg/dL.
6. Duration of disease since diagnosis < 3 years.
7. Negative stool culture, Clostridium Difficile Toxin from current flare.

Exclusion Criteria:

1. Duration of disease since diagnosis > 3 years.
2. Positive stool culture or O&P last 30 days.
3. Presence of clostridium difficile toxin in stool.
4. Azithromycin or Metronidazole allergy or known intolerance.
5. Diagnosis of IBD -U.
6. Presence of macroscopic disease involving the proximal ileum or jejunum (L4b).
7. Continuous macroscopic disease of the colon appearing as typical ulcerative colitis and Crohns diagnosed only by focality or granuloma on biopsies.
8. Presence of extraintestinal manifestations (such as arthritis, uveitis, or sclerosing cholangitis).Apthous lesions of mouth can be included.
9. Presence of fibrostenotic disease (strictures with prestenotic dilatation).
10. Presence of penetrating disease (fistulas or abscess).
11. Presence of current perianal disease defined as fistula or abscess.
12. Patients receiving concurrent corticosteroids or biologics.
13. Patients who have received steroids in the past 14 days.
14. Immune deficiency (CGD, GSD1, IL10R etc).
15. Known allergy or intolerance to any of the study medications.
16. Concurrent diseases such as hepatitis, ALT >2 times UNL, renal failure.
17. Pregnancy.
18. Patients with known heart disease.
19. Prolonged QTc by E.C.G at baseline.
20. Patient after surgical resection.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2012-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Response rate at 8 weeks defined as a drop in PCDAI (Pediatric Crohn's Disease Activity Index ) of at least 12.5 points (or remission without steroids, intention to treat principle) | 8 weeks

SECONDARY OUTCOMES:
Normalization of CRP ( CRP ≤0.5 mg/dL). | At week 8
Fecal calprotectin at 8 weeks . | 8 weeks
Remission at week 8 | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Arie Levine, MD, Study Chair — Pediatric Gastroenterology and Nutrition Unit, The E. Wolfson MC, Tel-Aviv University, Holon, Israel; Dan Turner, MD, PhD, Study Director — Pediatric Gastroenterology and Nutrition Unit, The Hebrew University of Jerusalem, Shaare Zedek MC, Jerusalem, Israel; Athos Bousvaros, MD, Study Director — Bostons Childrens Hospital; Michal Kori, MD, Principal Investigator — Kaplan Medical Center; Ron Shaoul, MD, Principal Investigator — Rambam Health Care Campus; Eyath Wine, MD, Principal Investigator — Women and Children's Health Research Institute, University of Alberta, Edmonton; Jorge Amil Dias, MD, Principal Investigator — Hospital S. Joao, Porto, Porpugal; Gigi Wauters Veereman, MD, Principal Investigator — Pedigastro, Antwerpen, Belgium; Malgorzata Margaret Sladek, MD, PhD, Principal Investigator — Polish-American Children's Hospital; Richard Russell, MD, Principal Investigator — Yorkhill Hospital, Glasgow, Scotland; Johanna C. (Hankje), Escher, MD PhD, Principal Investigator — Erasmus MC-Sophia Children's Hospital
Locations (1):
- The E. Wolfson.Medical Center, Holon, Israel

REFERENCES:
- [Derived] Levine A, Kori M, Kierkus J, Sigall Boneh R, Sladek M, Escher JC, Wine E, Yerushalmi B, Amil Dias J, Shaoul R, Veereman Wauters G, Boaz M, Abitbol G, Bousvaros A, Turner D. Azithromycin and metronidazole versus metronidazole-based therapy for the induction of remission in mild to moderate paediatric Crohn's disease : a randomised controlled trial. Gut. 2019 Feb;68(2):239-247. doi: 10.1136/gutjnl-2017-315199. Epub 2018 Feb 2. PMID 29420227